CLINICAL TRIAL: NCT01272232
Title: Effect of Liraglutide on Body Weight in Overweight or Obese Subjects With Type 2 Diabetes: A 56 Week Randomised, Double-blind, Placebo-controlled, Three Armed Parallel Group, Multi-centre, Multinational Trial With a 12 Week Observational Follow-up Period
Brief Title: Effect of Liraglutide on Body Weight in Overweight or Obese Subjects With Type 2 Diabetes: SCALE™ - Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-1922; 2008-002199-88 (EudraCT Number); U1111-1118-7963 (Other: WHO)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lira 3.0 mg (Experimental)
  Interventions: Drug: liraglutide
- Lira 1.8 mg (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Experimental)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Liraglutide 3.0 mg for subcutaneous (under the skin) injection once daily for 56 weeks.
  Arms: Lira 3.0 mg
Drug: liraglutide — Liraglutide 1.8 mg for subcutaneous (under the skin) injection once daily for 56 weeks.
  Arms: Lira 1.8 mg
Drug: placebo — Liraglutide placebo of either 3.0 mg or 1.8 mg for subcutaneous (under the skin) injection once daily for 56 weeks.
  Arms: Placebo

SUMMARY:
This trial is conducted in Africa, Asia, Europe and the United States of America (USA).

The aim of this trial is to investigate the potential of liraglutide to induce and maintain weight loss in overweight or obese subjects with type 2 diabetes. Treatment will be added onto subject's pre-trial background diabetes treatment of either diet and exercise only or single compound oral antidiabetic drug (OAD) treatment (metformin, sulphonylurea [SU] or glitazone) or combination OAD treatment (metformin, sulphonylurea or glitazone). The duration of the trial will be 56 weeks followed by a 12 week observational follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Subjects diagnosed with type 2 diabetes and treated with either diet and exercise alone, metformin, sulphonylurea, glitazone as single agent therapy or a combination of the previously mentioned compounds
* HbA1c 7.0-10.0% (both inclusive)
* Body Mass Index (BMI) at least 27.0 kg/m^2
* Stable body weight
* Preceding failed dietary effort

Exclusion Criteria:

* Treatment with glucagon-like peptide-1 (GLP-1) receptor agonists, dipeptidyl peptidase-4 (DPP-4) inhibitors or insulin within the last 3 months
* Known proliferative retinopathy or maculopathy
* History of acute or chronic pancreatitis
* Obesity induced by drug treatment
* Use of approved weight lowering pharmacotherapy
* Previous surgical treatment of obesity
* History of major depressive disorder or suicide attempt
* Uncontrolled hypertension (systolic blood pressure above or equal to 160 mmHg and/or diastolic blood pressure above or equal to 100 mmHg)
* Screening calcitonin of 50 ng/L or above
* Familial or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC)
* Personal history of non-familial medullary thyroid carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 846 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2013-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (144):
- United States (60):
  - Novo Nordisk Investigational Site, Vestavia Hills, Alabama
  - Novo Nordisk Investigational Site, Peoria, Arizona
  - Novo Nordisk Investigational Site, Jonesboro, Arkansas
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Arvada, Colorado
  - Novo Nordisk Investigational Site, Brooksville, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Columbus, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Columbia, Maryland
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Southfield, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Endwell, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Hickory, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Salisbury, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Anderson, South Carolina
  - Novo Nordisk Investigational Site, Moncks Corner, South Carolina
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
- France (8):
  - Novo Nordisk Investigational Site, Bondy
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Pointe à Pitre
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (10):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Gebhardshain
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Heidelberg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Schkeuditz
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Wangen
- India (5):
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Pune
  - Novo Nordisk Investigational Site, Thriruvananthapuram
- Israel (5):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Rishon LeZiyyon
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Italy (9):
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Chieti Scalo
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Forlì
  - Novo Nordisk Investigational Site, Latina
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Perugia
  - Novo Nordisk Investigational Site, Pistoia
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- South Africa (8):
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Lenasia, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Brits, North West
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- Spain (5):
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Partida de Bacarot
  - Novo Nordisk Investigational Site, Seville
- Sweden (7):
  - Novo Nordisk Investigational Site, Ängelholm
  - Novo Nordisk Investigational Site, Dalby
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Luleå
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Stockholm
- Taiwan (3):
  - Novo Nordisk Investigational Site, Taichung
  - Novo Nordisk Investigational Site, Tainan
  - Novo Nordisk Investigational Site, Taoyuan District
- Turkey (Türkiye) (6):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Gaziantep
  - Novo Nordisk Investigational Site, Hatay
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
  - Novo Nordisk Investigational Site, Kahramanmaraş
- United Kingdom (17):
  - Novo Nordisk Investigational Site, Airdrie
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Bexhill-on-Sea
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Chester
  - Novo Nordisk Investigational Site, Darlington
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Middlesbrough
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Rotherham
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Truro

REFERENCES:
- [Background] le Roux C, Aroda V, Hemmingsson J, Cancino AP, Christensen R, Pi-Sunyer X. Comparison of Efficacy and Safety of Liraglutide 3.0 mg in Individuals with BMI above and below 35 kg/m(2): A Post-hoc Analysis. Obes Facts. 2017;10(6):531-544. doi: 10.1159/000478099. Epub 2017 Nov 17. PMID 29145215
- [Result] Overgaard RV, Petri KC, Jacobsen LV, Jensen CB. Liraglutide 3.0 mg for Weight Management: A Population Pharmacokinetic Analysis. Clin Pharmacokinet. 2016 Nov;55(11):1413-1422. doi: 10.1007/s40262-016-0410-7. PMID 27193270
- [Result] O'Neil PM, Garvey WT, Gonzalez-Campoy JM, Mora P, Ortiz RV, Guerrero G, Claudius B, Pi-Sunyer X; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. EFFECTS OF LIRAGLUTIDE 3.0 MG ON WEIGHT AND RISK FACTORS IN HISPANIC VERSUS NON-HIPANIC POPULATIONS: SUBGROUP ANALYSIS FROM SCALE RANDOMIZED TRIALS. Endocr Pract. 2016 Nov;22(11):1277-1287. doi: 10.4158/EP151181.OR. Epub 2016 Aug 2. PMID 27482610
- [Result] Fujioka K, O'Neil PM, Davies M, Greenway F, C W Lau D, Claudius B, Skjoth TV, Bjorn Jensen C, P H Wilding J. Early Weight Loss with Liraglutide 3.0 mg Predicts 1-Year Weight Loss and is Associated with Improvements in Clinical Markers. Obesity (Silver Spring). 2016 Nov;24(11):2278-2288. doi: 10.1002/oby.21629. PMID 27804269
- [Result] Bays H, Pi-Sunyer X, Hemmingsson JU, Claudius B, Jensen CB, Van Gaal L. Liraglutide 3.0 mg for weight management: weight-loss dependent and independent effects. Curr Med Res Opin. 2017 Feb;33(2):225-229. doi: 10.1080/03007995.2016.1251892. Epub 2016 Nov 6. PMID 27817208
- [Result] Ard J, Cannon A, Lewis CE, Lofton H, Vang Skjoth T, Stevenin B, Pi-Sunyer X. Efficacy and safety of liraglutide 3.0 mg for weight management are similar across races: subgroup analysis across the SCALE and phase II randomized trials. Diabetes Obes Metab. 2016 Apr;18(4):430-5. doi: 10.1111/dom.12632. Epub 2016 Feb 11. PMID 26744025
- [Result] Wilding JP, Overgaard RV, Jacobsen LV, Jensen CB, le Roux CW. Exposure-response analyses of liraglutide 3.0 mg for weight management. Diabetes Obes Metab. 2016 May;18(5):491-9. doi: 10.1111/dom.12639. Epub 2016 Mar 1. PMID 26833744
- [Result] Davies MJ, Bergenstal R, Bode B, Kushner RF, Lewin A, Skjoth TV, Andreasen AH, Jensen CB, DeFronzo RA; NN8022-1922 Study Group. Efficacy of Liraglutide for Weight Loss Among Patients With Type 2 Diabetes: The SCALE Diabetes Randomized Clinical Trial. JAMA. 2015 Aug 18;314(7):687-99. doi: 10.1001/jama.2015.9676. PMID 26284720
- [Result] McEvoy BW. Missing data in clinical trials for weight management. J Biopharm Stat. 2016;26(1):30-6. doi: 10.1080/10543406.2015.1094814. PMID 26418188
- [Result] Steinberg WM, Rosenstock J, Wadden TA, Donsmark M, Jensen CB, DeVries JH. Impact of Liraglutide on Amylase, Lipase, and Acute Pancreatitis in Participants With Overweight/Obesity and Normoglycemia, Prediabetes, or Type 2 Diabetes: Secondary Analyses of Pooled Data From the SCALE Clinical Development Program. Diabetes Care. 2017 Jul;40(7):839-848. doi: 10.2337/dc16-2684. Epub 2017 May 4. PMID 28473337
- [Result] von Scholten BJ, Davies MJ, Persson F, Hansen TW, Madsbad S, Endahl L, Jepsen CH, Rossing P. Effect of weight reductions on estimated kidney function: Post-hoc analysis of two randomized trials. J Diabetes Complications. 2017 Jul;31(7):1164-1168. doi: 10.1016/j.jdiacomp.2017.04.003. Epub 2017 Apr 11. PMID 28462892
- [Result] O'Neil PM, Aroda VR, Astrup A, Kushner R, Lau DCW, Wadden TA, Brett J, Cancino AP, Wilding JPH; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Neuropsychiatric safety with liraglutide 3.0 mg for weight management: Results from randomized controlled phase 2 and 3a trials. Diabetes Obes Metab. 2017 Nov;19(11):1529-1536. doi: 10.1111/dom.12963. Epub 2017 Jul 21. PMID 28386912
- [Result] Davies MJ, Aronne LJ, Caterson ID, Thomsen AB, Jacobsen PB, Marso SP; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Liraglutide and cardiovascular outcomes in adults with overweight or obesity: A post hoc analysis from SCALE randomized controlled trials. Diabetes Obes Metab. 2018 Mar;20(3):734-739. doi: 10.1111/dom.13125. Epub 2017 Nov 1. PMID 28950422
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 126 sites in 9 countries participated: France (7), Germany (10), Israel (5), South Africa (6), Spain (8), Sweden (5), Turkey (3), United Kingdom (15), United States (67).
Pre-assignment Details: If eligible based on screened assessments, subjects were randomised to 1 of the 3 treatment arms in a 2:1:1 manner (liraglutide 3.0 mg, liraglutide 1.8 mg and placebo, respectively).
Groups:
- Liraglutide 3.0 mg: Exposed subjects received 56 weeks of once-daily subcutaneous (s.c.) injections with liraglutide, titrated from a starting dose of 0.6 mg in weekly increments of 0.6 mg to the target dose of 3.0 mg. In the 12-week follow-up period, treatment was discontinued. In addition to liraglutide 3.0 mg treatment, subjects were instructed to follow a hypocaloric diet and an exercise programme. Pre-trial treatment with metformin, glitazone or sulphonorylureas (SU) was continued throughout the trial (open-label) at unchanged dose, expect for SU that was reduced by 50%.
- Liraglutide 1.8 mg: Exposed subjects received 56 weeks of once-daily subcutaneous (s.c.) injections with liraglutide, titrated from a starting dose of 0.6 mg in weekly increments of 0.6 mg to the target dose of 1.8 mg. In the 12-week follow-up period, treatment was discontinued. In addition to liraglutide 1.8 mg treatment, subjects were instructed to follow a hypocaloric diet and an exercise programme. Pre-trial treatment with metformin, glitazone or sulphonorylureas (SU) was continued throughout the trial (open-label) at unchanged dose, expect for SU that was reduced by 50%.
- Liraglutide Placebo: Exposed subjects received 56 weeks of once-daily subcutaneous (s.c.) injections with liraglutide placebo. In the 12-week follow-up period, treatment was discontinued. In addition to placebo treatment, subjects were instructed to follow a hypocaloric diet and an exercise programme. Pre-trial treatment with metformin, glitazone or sulphonorylureas (SU) was continued throughout the trial (open-label) at unchanged dose, expect for SU that was reduced by 50%.
Period: Weeks 0-56
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Started | 423 | 211 | 212
Exposed | 422 (1 subject dropped out after randomisation and before exposure to trial drug.) | 210 (1 subject dropped out after randomisation and before exposure to trial drug.) | 212
Completed | 324 | 164 | 140
Not Completed | 99 | 47 | 72
Not completed — Adverse Event | 39 | 18 | 7
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Protocol Violation | 12 | 8 | 13
Not completed — Withdrawal criteria | 32 | 14 | 37
Not completed — Unclassified | 16 | 7 | 12
Period: Off Drug Follow-up Period (Weeks 56-68)
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Started | 324 | 164 | 140
Completed | 310 | 154 | 135
Not Completed | 14 | 10 | 5
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal criteria | 9 | 7 | 4
Not completed — Unclassified | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo | Total
Number analyzed (Participants) | 423 | 211 | 212 | 846
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (10.8) | 54.9 (10.7) | 54.7 (9.8) | 54.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 103 | 115 | 421
  Male | 220 | 108 | 97 | 425
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 17 | 24 | 87
  Not Hispanic or Latino | 375 | 194 | 187 | 756
  Unknown or Not Reported | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 0 | 4
  Asian | 11 | 4 | 4 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 44 | 27 | 27 | 98
  White | 353 | 177 | 175 | 705
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 3 | 6 | 20
Age group [Number; unit: participants]
  18- < 40 years | 38 | 15 | 13 | 66
  40- < 65 years | 300 | 162 | 161 | 623
  65- < 75 years | 74 | 32 | 36 | 142
  >= 75 years | 11 | 2 | 2 | 15
Fasting body weight [Mean (Standard Deviation); unit: kg] — Weight was recorded to the nearest 0.1 kg for a subject in the fasting state with an empty bladder, without shoes and only wearing light clothing. The same calibrated scale was used throughout the trial.
  kg | 105.7 (21.9) | 105.8 (21.0) | 106.5 (21.3) | 105.9 (21.5)
Height [Mean (Standard Deviation); unit: m] — Height was recorded without shoes.
  m | 1.69 (0.11) | 1.69 (0.10) | 1.69 (0.10) | 1.69 (0.10)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 37.1 (6.5) | 37.0 (6.9) | 37.4 (7.1) | 37.1 (6.8)
Body Mass Index (BMI) group [Number; unit: participants]
  25.0-29.9 kg/m^2 - pre-obese | 52 | 34 | 30 | 116
  30.0-34.9 kg/m^2 - obese class I | 139 | 62 | 59 | 260
  35.0-39.9 kg/m^2 - obese class II | 108 | 50 | 60 | 218
  >40.0 kg/m^2 - obese class III | 124 | 65 | 63 | 252
HbA1c (glycosylated haemoglobin) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] | 7.9 (0.8) | 8.0 (0.8) | 7.9 (0.8) | 7.9 (0.8)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] | 8.8 (1.9) | 8.9 (2.0) | 8.6 (1.8) | 8.8 (1.9)
Co-morbid hypertension [Number; unit: participants] — Presence or absence of untreated or treated hypertension
  participants
    Present | 293 | 148 | 145 | 586
    Absent | 130 | 63 | 67 | 260
Co-morbid dyslipidaemia [Number; unit: participants] — Presence or absence of untreated or treated dyslipidaemia
  participants
    Present | 295 | 143 | 126 | 564
    Absent | 128 | 68 | 86 | 282
Duration of diabetes [Mean (Standard Deviation); unit: years] | 7.54 (5.65) | 7.43 (5.16) | 6.71 (5.07) | 7.30 (5.39)

OUTCOME MEASURES:

1. Primary Outcome: Change (%) From Baseline in Body Weight (Fasting)
Description: Weight was recorded to the nearest 0.1 kg for a subject in the fasting state with an empty bladder, without shoes and only wearing light clothing. The same calibrated scale was used throughout the trial.
Time Frame: Week 0, week 56
Population: Last Observation Carried Forward (LOCF) data. Full analysis set, comprising all randomised subjects who had been exposed to at least 1 dose of trial product and with at least 1 post-randomisation assessment of any efficacy endpoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 412 | 204 | 211
percent change | -5.9 (5.5) | -4.6 (5.5) | -2.0 (4.3)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Liraglutide Placebo; The 3 co-primary endpoints (Outcome Measures 1, 2 and 3) were ranked (#1, 2, 3); hypotheses of no difference were tested in a hierarchical manner. Fixed factors: treatment, country, sex, background treatment, baseline HbA1c stratum, background treatment/HbA1c-stratum-interaction; covariate: baseline value; Test type: Superiority or Other; p < 0.0001, ANCOVA — Superiority was established only if all preceding hypotheses had been rejected. p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -3.97, 95% CI [-4.84 to -3.11]
Statistical Analysis 2: Comparison: Liraglutide 1.8 mg vs Liraglutide Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Treatment contrast = -2.62, 95% CI [-3.63 to -1.62]
Statistical Analysis 3: Comparison: Liraglutide 3.0 mg vs Liraglutide 1.8 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0024, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Treatment contrast = -1.35, 95% CI [-2.23 to -0.48]

2. Primary Outcome: Proportion of Subjects Losing at Least 5% of Baseline Body Weight
Description: as for outcome 1
Time Frame: at 56 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 412 | 204 | 211
percentage of subjects
  Yes | 49.9 | 35.6 | 13.8
  No | 50.1 | 64.4 | 86.2
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Liraglutide Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 6.81, 95% CI [4.34 to 10.68]
Statistical Analysis 2: Comparison: Liraglutide 1.8 mg vs Liraglutide Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.69, 95% CI [2.24 to 6.09]
Statistical Analysis 3: Comparison: Liraglutide 3.0 mg vs Liraglutide 1.8 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0008, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.84, 95% CI [1.29 to 2.64]

3. Primary Outcome: Proportion of Subjects Losing More Than 10% of Baseline Body Weight
Description: as for outcome 1
Time Frame: at 56 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 412 | 204 | 211
percentage of subjects
  Yes | 23.4 | 14.4 | 4.3
  No | 76.6 | 85.6 | 95.7
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Liraglutide Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.10, 95% CI [3.48 to 14.48]
Statistical Analysis 2: Comparison: Liraglutide 1.8 mg vs Liraglutide Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0008, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.84, 95% CI [1.75 to 8.41]
Statistical Analysis 3: Comparison: Liraglutide 3.0 mg vs Liraglutide 1.8 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0099, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.85, 95% CI [1.16 to 2.95]

4. Secondary Outcome: Change (%-Points) From Baseline in HbA1c (Glycosylated Haemoglobin A1c)
Description: Change in HbA1c (%-points) was calculated as the difference between the HbA1c (%) at Week 0 and Week 56.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage point change of HbA1c
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 412 | 204 | 211
percentage point change of HbA1c | -1.3 (0.9) | -1.1 (1.0) | -0.3 (0.9)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Liraglutide Placebo; Test of no difference. Fixed factors: treatment, country, sex, background treatment, baseline HbA1c stratum, background treatment/HbA1c-stratum-interaction; covariate: baseline value; Test type: Superiority or Other; p < 0.0001, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -0.93, 95% CI [-1.08 to -0.78]
Statistical Analysis 2: Comparison: Liraglutide 1.8 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -0.74, 95% CI [-0.91 to -0.57]
Statistical Analysis 3: Comparison: Liraglutide 3.0 mg vs Liraglutide 1.8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0125, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -0.19, 95% CI [-0.34 to -0.04]

5. Secondary Outcome: Proportion of Subjects Reaching Target HbA1c Below 7%
Time Frame: at 56 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 412 | 204 | 211
percentage of subjects
  Yes | 69.2 | 66.7 | 27.2
  No | 30.8 | 33.3 | 72.8
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p values are 2-sided; 5% pre-defined significance level; Odds Ratio (OR) = 8.79, 95% CI [5.74 to 13.4]
Statistical Analysis 2: Comparison: Liraglutide 1.8 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p values are 2-sided; 5% pre-defined significance level; Odds Ratio (OR) = 7.71, 95% CI [4.76 to 12.51]
Statistical Analysis 3: Comparison: Liraglutide 3.0 mg vs Liraglutide 1.8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.5319, Regression, Logistic — p values are 2-sided; 5% pre-defined significance level; Odds Ratio (OR) = 1.14, 95% CI [0.76 to 1.71]

6. Secondary Outcome: Proportion of Subjects Reaching Target HbA1c Below or Equal to 6.5%
Time Frame: at 56 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 412 | 204 | 211
percentage of subjects
  Yes | 56.5 | 45.6 | 15.0
  No | 43.5 | 54.4 | 85.0
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p values are 2-sided; 5% pre-defined significance level; Odds Ratio (OR) = 9.61, 95% CI [6.05 to 15.26]
Statistical Analysis 2: Comparison: Liraglutide 1.8 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p values are 2-sided; 5% pre-defined significance level; Odds Ratio (OR) = 5.98, 95% CI [3.59 to 9.97]
Statistical Analysis 3: Comparison: Liraglutide 3.0 mg vs Liraglutide 1.8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0142, Regression, Logistic — p values are 2-sided; 5% pre-defined significance level; Odds Ratio (OR) = 1.61, 95% CI [1.10 to 2.34]

7. Secondary Outcome: Change From Baseline in Waist Circumference
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 412 | 204 | 211
cm | -6.1 (6.5) | -4.8 (5.6) | -2.7 (5.4)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -3.22, 95% CI [-4.20 to -2.23]
Statistical Analysis 2: Comparison: Liraglutide 1.8 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0004, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -2.06, 95% CI [-3.20 to -0.92]
Statistical Analysis 3: Comparison: Liraglutide 3.0 mg vs Liraglutide 1.8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0224, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -1.16, 95% CI [-2.16 to -0.16]

8. Secondary Outcome: Change (%) From Baseline in Body Weight (Fasting)
Description: as for outcome 1
Time Frame: Week 0, week 68
Population: Full analysis set, comprising all randomised subjects who had been exposed to at least 1 dose of trial product and with at least 1 post-randomisation assessment of any efficacy endpoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 324 | 164 | 140
percent change | -4.7 (5.0) | -3.6 (5.7) | -2.7 (5.8)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -2.17, 95% CI [-3.32 to -1.02]
Statistical Analysis 2: Comparison: Liraglutide 1.8 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0725, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -1.20, 95% CI [-2.51 to 0.11]
Statistical Analysis 3: Comparison: Liraglutide 3.0 mg vs Liraglutide 1.8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0717, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -0.97, 95% CI [-2.02 to 0.09]

9. Secondary Outcome: Change (%) From Week 56 to 68 in Body Weight (Fasting)
Description: as for outcome 1
Time Frame: Week 56, week 68
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 324 | 164 | 140
percent change | 2.3 (2.9) | 2.0 (2.9) | -0.1 (2.2)

10. Secondary Outcome: Change From Baseline in Waist Circumference
Time Frame: Week 0, week 68
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 324 | 164 | 140
cm | -5.7 (6.3) | -4.4 (6.0) | -3.2 (6.8)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -2.49, 95% CI [-3.75 to -1.24]
Statistical Analysis 2: Comparison: Liraglutide 1.8 mg vs Liraglutide Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0457, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -1.47, 95% CI [-2.92 to -0.03]
Statistical Analysis 3: Comparison: Liraglutide 3.0 mg vs Liraglutide 1.8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0961, ANCOVA — p values are 2-sided; 5% pre-defined significance level; Treatment contrast = -1.02, 95% CI [-2.22 to 0.18]

11. Secondary Outcome: Change From Week 56 to 68 in Waist Circumference
Time Frame: Week 56, week 68
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 324 | 164 | 140
cm | 1.21 (3.94) | 1.02 (3.55) | -0.22 (3.23)

12. Secondary Outcome: Incidence of Hypoglycaemic Episodes
Description: Hypoglycaemic episodes were classified according to American Diabetes Association (ADA) definitions as well as to the Novo Nordisk definition of a minor hypoglycaemic event (blood glucose level below approximately 2.8 mmol/L [50 mg/dL] or plasma glucose level below 3.1 mmol/L [56 mg/dL]).
Time Frame: Weeks 0-56
Population: Safety analysis set, comprising all randomised subjects who had been exposed to at least one dose of trial product.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Number analyzed (Participants) | 422 | 210 | 212
Episodes/100 years of patient exposure
  Minor | 34 | 46 | 13
  ADA: Severe | 1 | 2 | 0
  ADA: Documented, symptomatic | 87 | 95 | 31
  ADA: Asymptomatic | 151 | 142 | 46
  ADA: Probable, symptomatic | 2 | 2 | 1
  ADA: Relative | 17 | 16 | 5
  ADA: Unclassifiable | 14 | 7 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for up to 68 weeks.
Description: Safety Analysis Set comprising all randomised subjects who had been exposed to at least one dose of trial product.
Arm/Group | Liraglutide 3.0 mg | Liraglutide 1.8 mg | Liraglutide Placebo
Serious Adverse Events (participants affected / at risk) | 37/422 | 18/210 | 13/212
Other Adverse Events (participants affected / at risk) | 361/422 | 173/210 | 164/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg (N=422) | Liraglutide 1.8 mg (N=210) | Liraglutide Placebo (N=212)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Meniere (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood calcitonin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Coronary revascularisation (Surgical and medical procedures) | 2 (2) | 0 (0) | 1 (2)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Nasal operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg (N=422) | Liraglutide 1.8 mg (N=210) | Liraglutide Placebo (N=212)
Abdominal distension (Gastrointestinal disorders) | 26 (32) | 10 (11) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 26 (34) | 4 (4) | 9 (9)
Abdominal pain upper (Gastrointestinal disorders) | 15 (21) | 14 (17) | 2 (2)
Constipation (Gastrointestinal disorders) | 68 (78) | 20 (24) | 13 (14)
Diarrhoea (Gastrointestinal disorders) | 108 (173) | 37 (50) | 27 (35)
Dyspepsia (Gastrointestinal disorders) | 47 (59) | 14 (16) | 5 (5)
Flatulence (Gastrointestinal disorders) | 22 (26) | 8 (8) | 4 (4)
Nausea (Gastrointestinal disorders) | 138 (208) | 66 (84) | 29 (34)
Vomiting (Gastrointestinal disorders) | 66 (113) | 21 (27) | 12 (14)
Fatigue (General disorders) | 35 (45) | 11 (11) | 7 (7)
Injection site haematoma (General disorders) | 19 (33) | 4 (4) | 12 (14)
Bronchitis (Infections and infestations) | 13 (14) | 12 (16) | 11 (15)
Influenza (Infections and infestations) | 22 (24) | 12 (14) | 15 (16)
Nasopharyngitis (Infections and infestations) | 88 (134) | 34 (46) | 41 (54)
Sinusitis (Infections and infestations) | 16 (19) | 15 (18) | 18 (22)
Upper respiratory tract infection (Infections and infestations) | 40 (49) | 23 (25) | 18 (19)
Urinary tract infection (Infections and infestations) | 19 (34) | 13 (17) | 12 (14)
Lipase increased (Investigations) | 50 (56) | 22 (26) | 14 (16)
Decreased appetite (Metabolism and nutrition disorders) | 40 (44) | 23 (23) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 187 (981) | 84 (429) | 59 (154)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (42) | 17 (25) | 12 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 42 (67) | 27 (36) | 20 (27)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 22 (24) | 9 (10) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (20) | 12 (13) | 10 (12)
Dizziness (Nervous system disorders) | 30 (39) | 10 (15) | 6 (7)
Headache (Nervous system disorders) | 66 (125) | 26 (42) | 29 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 12 (16) | 8 (9)
Hypertension (Vascular disorders) | 12 (12) | 7 (8) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right not to release data until specified milestones are available. This includes the right not to release interim results from clinical trials, as such results may lead to conclusions that are later proven incorrect. At the end of the trial, one or more manuscripts for publication will be prepared in collaboration between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to briefly postpone publication or communication to protect intellectual property.